CLINICAL TRIAL: NCT02655679
Title: A Randomized, Double-Blind, Vehicle-Controlled Ascending Multiple Dose and Clinical Proof-Of-Concept Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of VTP-38543 in Adult Patients With Mild to Moderate Atopic Dermatitis
Brief Title: An Ascending Multiple Dose Study of VTP-38543 in Adult Participants With Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vitae Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VTP-38543-001
Record Dates: First submitted 2016-01-11; First posted 2016-01-14 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Dermatitis, Atopic
Keywords: Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- VTP-38543 0.05% (Experimental): VTP-38543 0.05% administered topically every 12 hours for 28 days.
  Interventions: Drug: VTP-38543
- VTP-38543 0.15% (Experimental): VTP-38543 0.15% administered topically every 12 hours for 28 days.
  Interventions: Drug: VTP-38543
- Vehicle without Transcutol®P (Placebo Comparator): Vehicle without Transcutol®P administered topically every 12 hours for 28 days.
  Interventions: Other: Vehicle without Transcutol®P
- VTP-38543 1% (Experimental): VTP-38543 1% administered topically every 12 hours for 28 days.
  Interventions: Drug: VTP-38543
- Vehicle with Transcutol®P (Placebo Comparator): Vehicle with Transcutol®P administered topically every 12 hours for 28 days.
  Interventions: Other: Vehicle with Transcutol®P

INTERVENTIONS:
Drug: VTP-38543 — VTP-38543 topical cream
  Arms: VTP-38543 0.05%; VTP-38543 0.15%; VTP-38543 1%
Other: Vehicle with Transcutol®P — Vehicle matching VTP-38543 cream with Transcutol®P
  Other Names: Transcutol®P is Diethylene Glycol Monoethyl Ether, NF.
  Arms: Vehicle with Transcutol®P
Other: Vehicle without Transcutol®P — Vehicle matching VTP-38543 cream without Transcutol®P
  Other Names: Transcutol®P is Diethylene Glycol Monoethyl Ether, NF.
  Arms: Vehicle without Transcutol®P

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and preliminary clinical efficacy of VTP-38543 administered as a cream, twice-daily, for 28 days in otherwise healthy adult male and female participants with mild to moderate atopic dermatitis.

DETAILED DESCRIPTION:
This is a randomized, double-blind, vehicle-controlled study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and preliminary clinical efficacy of VTP-38543 following twice-daily, every twelve hours (Q12h) administration for 28 days in otherwise healthy adult male and female participants with mild to moderate atopic dermatitis.

Evaluation of three ascending doses in three dose panels is planned for this trial. Dose Panel 1 (VTP-38543 0.05%) and Panel 2 (VTP-38543 0.15%) will each enroll 30 participants and randomize 20 to VTP-38543 and 10 to matching vehicle control (Vehicle without Transcutol®P). Dose Panel 3 (VTP-38543 1%) will enroll 40 participants and randomize 20 to VTP-38543 and 20 to matching vehicle control (Vehicle with Transcutol®P). A total of approximately 100 participants will participate in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate atopic dermatitis with a minimum of 3 to a maximum of 15% body surface area (BSA) involvement
* Investigator Global Assessments (IGA) score of 2 or 3
* Body Mass Index (BMI) = 18 - 35 kg/m^2
* Negative Pregnancy test for females

Exclusion Criteria:

* Treatment for atopic dermatitis with systemic medications, topical agents, and parenteral biological/monoclonal antibody agents, within specific time period prior to dosing.
* Organ dysfunction or any clinically significant deviation from normal in vital signs, physical examinations, labs, and Electrocardiogram (ECG) findings
* Major surgery within 3 months of Screening
* Use of prescription drugs, sedative antihistamine, medical devices for treatment of atopic dermatitis (AD), and topical products containing urea and/or ceramides within 14 prior to dosing
* Excessive sun exposures, use of tanning booths or other ultraviolet (UV) light sources 4 weeks prior to dosing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2016-09-09 (Actual); Study Completion 2016-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christy Harutunian, Study Director — Allergan
Locations (12):
- United States (5):
  - Dundee Dermatology, West Dundee, Illinois
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Skin Specialty Dermatology, New York, New York
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Paddington Testing Company, Inc, Philadelphia, Pennsylvania
- Canada (7):
  - Kirk Barber Research, Calgary, Alberta
  - Stratica Medical Inc, Edmonton, Alberta
  - Lynderm Research Inc, Markham, Ontario
  - The Center for Dermatology / Institution, Richmond Hill, Ontario
  - Windsor Clinical Research Inc, Windsor, Ontario
  - Dr Isabelle Delorme Inc, Drummondville, Quebec
  - Innovaderm Research, Montreal, Quebec

REFERENCES:
- [Derived] Czarnowicki T, Dohlman AB, Malik K, Antonini D, Bissonnette R, Chan TC, Zhou L, Wen HC, Estrada Y, Xu H, Bryson C, Shen J, Lala D, Ma'ayan A, McGeehan G, Gregg R, Guttman-Yassky E. Effect of short-term liver X receptor activation on epidermal barrier features in mild to moderate atopic dermatitis: A randomized controlled trial. Ann Allergy Asthma Immunol. 2018 Jun;120(6):631-640.e11. doi: 10.1016/j.anai.2018.03.013. Epub 2018 Mar 19. PMID 29567358

RESULTS

PARTICIPANT FLOW:
Groups:
- VTP- 38543 0.05%: VTP-38543 0.05% administered topically every 12 hours for 28 days.
- VTP- 38543 0.15%: VTP-38543 0.15% administered topically every 12 hours for 28 days.
Period: Overall Study
Arm/Group | VTP- 38543 0.05% | VTP- 38543 0.15% | Vehicle Without Transcutol®P | VTP-38543 1% | Vehicle With Transcutol®P
Started | 21 | 19 | 20 | 24 | 20
Received Study Drug (Safety Population) | 20 | 19 | 20 | 24 | 20
Completed | 18 | 16 | 19 | 20 | 19
Not Completed | 3 | 3 | 1 | 4 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 3 | 1
Not completed — Inability to Comply with the Protocol | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1 | 0
Not completed — Other Miscellaneous Reasons | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included randomized participants who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | VTP- 38543 0.05% | VTP- 38543 0.15% | Vehicle Without Transcutol®P | VTP-38543 1% | Vehicle With Transcutol®P | Total
Number analyzed (Participants) | 20 | 19 | 20 | 24 | 20 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (15.79) | 36.8 (13.39) | 30.8 (11.59) | 35.7 (10.51) | 30.9 (11.73) | 34.1 (12.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 8 | 14 | 9 | 55
  Male | 7 | 8 | 12 | 10 | 11 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events (AEs)
Description: An Adverse Event is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The number of participants with AEs related to treatment are reported.
Time Frame: Baseline (Day 0) to Day 35
Population: Safety population included randomized participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | VTP-38543 0.05% | VTP-38543 0.15% | Vehicle Without Transcutol®P | VTP-38543 1% | Vehicle With Transcutol®P
Number analyzed (Participants) | 20 | 19 | 20 | 24 | 20
Participants | 1 | 3 | 2 | 6 | 2

2. Primary Outcome: Number of Participants With Clinically Significant Changes in Clinical Laboratory Values
Description: Clinical Laboratory tests included chemistry, hematology and urinalysis tests collected during the study. The investigator determined if the changes in laboratory results were clinically significant.
Time Frame: Baseline (Day 0) to Day 35
Population: Safety population included randomized participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | VTP-38543 0.05% | VTP-38543 0.15% | Vehicle Without Transcutol®P | VTP-38543 1% | Vehicle With Transcutol®P
Number analyzed (Participants) | 20 | 19 | 20 | 24 | 20
Participants | 0 | 1 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Vital signs included blood pressure, pulse, respiration rate and body temperature. The investigator determined if the changes in vital sign results were clinically significant.
Time Frame: Baseline (Day 0) to Day 35
Population: Safety population included randomized participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | VTP-38543 0.05% | VTP-38543 0.15% | Vehicle Without Transcutol®P | VTP-38543 1% | Vehicle With Transcutol®P
Number analyzed (Participants) | 20 | 19 | 20 | 24 | 20
Participants | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Values
Description: A standard 12-lead ECG was performed. The investigator determined if the changes in ECG results were clinically significant.
Time Frame: Baseline (Day 0) to Day 35
Population: Safety population included randomized participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | VTP-38543 0.05% | VTP-38543 0.15% | Vehicle Without Transcutol®P | VTP-38543 1% | Vehicle With Transcutol®P
Number analyzed (Participants) | 20 | 19 | 20 | 24 | 20
Participants | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Maximum Plasma Concentration (Cmax) for VTP-38543-001
Time Frame: Day 0 (pre-dose, 1, 2, 4, 6, 9, and 12 hours post first dose), and Day 27 (pre-dose, 1, 2, 4, 6, 9, 12, 24, 48, and 72 hours post last dose)
Population: Pharmacokinetic (PK) population included all participants with available plasma concentration data with profiles adequate to determine PK parameters. Number analyzed is the number of participants with serial sampling data available at the given timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | VTP-38543 0.05% | VTP-38543 0.15% | VTP-38543 1%
Number analyzed (Participants) | 8 | 8 | 8
ng/mL
  Day 0: number analyzed (Participants) | 6 | 4 | 6
  Day 0 | 0.546 (1.16) | 0.221 (0.175) | 2.34 (3.29)
  Day 27: number analyzed (Participants) | 5 | 4 | 4
  Day 27 | 2.81 (5.35) | 2.28 (1.68) | 13.4 (12.7)

6. Secondary Outcome: Time to Maximum Plasma Concentrations (Tmax) for VTP-38543
Time Frame: as for outcome 5
Population: PK population included all participants with available plasma concentration data with profiles adequate to determine PK parameters. Number analyzed is the number of participants with serial sampling data available at the given timepoint.
Measure: Median (Full Range); unit: hour
Arm/Group | VTP-38543 0.05% | VTP-38543 0.15% | VTP-38543 1%
Number analyzed (Participants) | 8 | 8 | 8
hour
  Day 0: number analyzed (Participants) | 6 | 4 | 6
  Day 0 | 5.5 [2 to 9] | 9 [2 to 9] | 4 [2 to 9]
  Day 27: number analyzed (Participants) | 5 | 4 | 4
  Day 27 | 1 [0 to 4] | 6.5 [2 to 24] | 4 [4 to 9]

7. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve, From Time 0 to the Last Measurable Concentration (AUClast) for VTP-38543
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | VTP-38543 0.05% | VTP-38543 0.15% | VTP-38543 1%
Number analyzed (Participants) | 8 | 8 | 8
ng*hr/mL
  Day 0: number analyzed (Participants) | 6 | 4 | 6
  Day 0 | 2.27 (4.23) | 1.35 (1.41) | 20.0 (28.2)
  Day 27: number analyzed (Participants) | 5 | 4 | 4
  Day 27 | 129 (257) | 104 (77.5) | 720 (798)

8. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve, From Time 0 to 12 Hours (AUC0-12hr) for VTP-38543
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | VTP-38543 0.05% | VTP-38543 0.15% | VTP-38543 1%
Number analyzed (Participants) | 8 | 8 | 8
ng*hr/mL
  Day 0: number analyzed (Participants) | 6 | 4 | 6
  Day 0 | 2.27 (4.23) | 1.35 (1.41) | 20.0 (28.2)
  Day 27: number analyzed (Participants) | 5 | 4 | 4
  Day 27 | 23.6 (44.8) | 22.2 (18.2) | 144 (144)

9. Secondary Outcome: Elimination Half-life (t½) for VTP-38543
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | VTP-38543 0.05% | VTP-38543 0.15% | VTP-38543 1%
Number analyzed (Participants) | 8 | 8 | 8
hour
  Day 0: number analyzed (Participants) | 6 | 4 | 6
  Day 0 | NA (NA) — t1/2 was not achieved at Day 0. | NA (NA) — t1/2 was not achieved at Day 0. | NA (NA) — t1/2 was not achieved at Day 0.
  Day 27: number analyzed (Participants) | 5 | 4 | 4
  Day 27 | 58.6 (14.5) | 47.2 (12.2) | 246 (349)

10. Secondary Outcome: Percentage Change From Baseline in Total Body Surface Area (BSA)
Description: Percent BSA was estimated using the palmar surface of the participant's hand up to the proximal interphalangeal joint, including the thumb, to approximate 1% of the participant's BSA. The overall BSA affected by atopic dermatitis was evaluated from 0 to 100% and divided by 5 for a maximum of 20. A negative percentage change indicates improvement.
Time Frame: Baseline (Day 0) to Day 28
Population: Modified intent-to-treat (mITT) population included all participants who were randomized and who received at least one dose of study medication and with a Baseline and Day 28 value for efficacy parameters.
Measure: Mean (Standard Deviation); unit: percentage change in total BSA
Arm/Group | VTP-38543 0.05% | VTP-38543 0.15% | Vehicle Without Transcutol®P | VTP-38543 1% | Vehicle With Transcutol®P
Number analyzed (Participants) | 17 | 16 | 18 | 19 | 19
percentage change in total BSA | -39.09 (29.233) | -9.46 (52.978) | -17.39 (55.588) | -9.44 (48.063) | -28.51 (29.398)

11. Secondary Outcome: Percentage Change From Baseline in Investigator Global Assessments (IGA) Score
Description: The investigator assessed the participant's atopic dermatitis using the 5-point IGA where 0=clear (Minor, residual discoloration, no erythema or induration/papulation, no oozing/crusting) to 4=Severe disease (Deep/bright red erythema with severe induration/papulation with oozing/crusting). A negative percentage change indicates improvement.
Time Frame: Baseline (Day 0) to Day 28
Population: mITT population included all participants who were randomized and who received at least one dose of study medication and with a Baseline and Day 28 value for efficacy parameters.
Measure: Mean (Standard Deviation); unit: percentage change in IGA score
Arm/Group | VTP-38543 0.05% | VTP-38543 0.15% | Vehicle Without Transcutol®P | VTP-38543 1% | Vehicle With Transcutol®P
Number analyzed (Participants) | 17 | 16 | 18 | 19 | 19
percentage change in IGA score | -12.7 (25.36) | -16.7 (34.96) | -19.4 (32.46) | -6.1 (34.79) | -13.2 (20.47)

12. Secondary Outcome: Percentage Change From Baseline in Scoring Atopic Dermatitis (SCORAD) Score
Description: The investigator assessed severity of atopic dermatitis (AD) using scoring atopic dermatitis (SCORAD) score obtained from different individual scales. 6-items: erythema, edema/papulation, oozing/crusts, excoriation, lichenification, and dryness were graded on a 4-point scale where 0=Absent to 3=Severe. The individual scores were added together to get a score of 0 to 18 that was multiplied by 3.5 for a score of 0 to 63. The overall BSA affected by AD (0 to 100 %) was divided by 5 for a score 0 to 20. The participant used a 10-point Visual Analog Scale (VAS) to evaluate loss of sleep and the occurrence of pruritus averaged over the last 3 days where 0=None to Worst Imaginable. The sum of the 2 VAS scores was 0 to 20. The above measures were added together for a total possible SCORAD score of 0 (best) to 103 (worst). A negative percentage change indicates improvement.
Time Frame: Baseline (Day 0) to Day 28
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage change in SCORAD score
Arm/Group | VTP-38543 0.05% | VTP-38543 0.15% | Vehicle Without Transcutol®P | VTP-38543 1% | Vehicle With Transcutol®P
Number analyzed (Participants) | 17 | 16 | 18 | 19 | 19
percentage change in SCORAD score | -23.473 (30.1085) | -17.300 (34.7270) | -24.453 (35.6572) | -14.483 (32.2743) | -18.630 (26.0370)

13. Secondary Outcome: Percentage Change From Baseline Eczema Area and Severity Index (EASI)
Description: The investigator assessed four body regions: Head and neck, Upper extremities, Trunk including axillae and groin, and Lower extremities including buttocks. Each body region was scored based on BSA where 0=No involvement to 6=90-100%. Each body region was assessed for erythema, infiltration/papulation, excoriation and lichenification using a 4-point scale where 0=None to 3=Severe. EASI total score was determined by combining the individual scores for each of the 4 body regions. The total for each region was calculated by [erythema + infiltration+ excoriation + lichenification * area involvement * a constant (constants Head and Neck=0.1, Upper Limbs=0.2, Trunk=0.3, Lower Limbs=0.4)]. The EASI total score was determined by combining the individual scores for each of the 4 body regions for a total possible score of 0 (best) to 72 (worst). A negative percentage change indicates improvement.
Time Frame: Baseline (Day 0) to Day 28
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage change in EASI
Arm/Group | VTP-38543 0.05% | VTP-38543 0.15% | Vehicle Without Transcutol®P | VTP-38543 1% | Vehicle With Transcutol®P
Number analyzed (Participants) | 17 | 16 | 18 | 19 | 19
percentage change in EASI | -36.26 (29.832) | -9.16 (66.519) | -26.99 (46.549) | -12.52 (58.819) | -27.10 (36.323)

14. Secondary Outcome: Percentage Change From Baseline in Pruritus VAS Score
Description: The participant used a 10-point VAS to assess the occurrence of pruritus (itchy skin) over the last 3 days where 0= None to 10=Worst Imaginable for a total possible score of 0 to 10. A negative percentage change indicates improvement.
Time Frame: Baseline (Day 0) to Day 28
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage change in pruritis VAS score
Arm/Group | VTP-38543 0.05% | VTP-38543 0.15% | Vehicle Without Transcutol®P | VTP-38543 1% | Vehicle With Transcutol®P
Number analyzed (Participants) | 17 | 16 | 18 | 19 | 19
percentage change in pruritis VAS score | 4.20 (112.105) | -20.07 (48.771) | -26.75 (47.715) | -25.80 (42.232) | -34.68 (54.612)

15. Secondary Outcome: Percentage Change From Baseline in VAS Sleep Score
Description: The participant used a 10-point VAS to evaluate loss of sleep averaged over the last 3 days where 0= None to 10=Worst imaginable for a total possible score of 0 to 10. A negative percentage change indicates improvement.
Time Frame: Baseline (Day 0) to Day 28
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage change in VAS sleep score
Arm/Group | VTP-38543 0.05% | VTP-38543 0.15% | Vehicle Without Transcutol®P | VTP-38543 1% | Vehicle With Transcutol®P
Number analyzed (Participants) | 15 | 13 | 15 | 18 | 13
percentage change in VAS sleep score | -29.40 (61.845) | -19.74 (78.382) | 2.73 (113.782) | -29.98 (53.672) | -30.85 (39.259)

ADVERSE EVENTS:
Time Frame: First dose of study drug to the last visit (Up to Day 35)
Description: Safety population, all randomized participants who received at least one dose of study medication, was used to determine the number of participants for Serious Adverse Events and Other Adverse Events.
Arm/Group | VTP- 38543 0.05% | VTP- 38543 0.15% | Vehicle Without Transcutol®P | VTP-38543 1% | Vehicle With Transcutol®P
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19 | 0/20 | 0/24 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/20 | 0/24 | 0/20
Other Adverse Events (participants affected / at risk) | 10/20 | 12/19 | 12/20 | 8/24 | 6/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VTP- 38543 0.05% (N=20) | VTP- 38543 0.15% (N=19) | Vehicle Without Transcutol®P (N=20) | VTP-38543 1% (N=24) | Vehicle With Transcutol®P (N=20)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Tooth impacted (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Application site pain (General disorders) | 1 | 1 | 1 | 3 | 1
Application site pruritus (General disorders) | 0 | 1 | 1 | 1 | 0
Administration site pruritus (General disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 2 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 3 | 3 | 1 | 0
Application site reaction (General disorders) | 0 | 0 | 0 | 2 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.